CLINICAL TRIAL: NCT06798883
Title: Perioperative Respiratory Support and Postoperative Outcomes: Russian National Epidemiological Study "RuVent-A"
Brief Title: Perioperative Respiratory Support and Postoperative Outcomes
Acronym: RuVent-A
Status: Not yet recruiting | Type: Observational
Sponsor: Russian Federation of Anesthesiologists and Reanimatologists (Other)
Responsible Party: Sponsor
Other Study IDs: FARCT0006
Record Dates: First submitted 2025-01-22; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Respiratory Complications
Keywords: anesthesia; respiratory support; complications; mechanical ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the methodology and parameters of perioperative respiratory support (RS) and the frequency of postoperative pulmonary complications (PPCs) in the Russian Federation. The study will analyze respiratory support strategies, equipment availability, and their correlation with PPC outcomes in surgical patients.

DETAILED DESCRIPTION:
Globally, around 230 million surgical procedures requiring general anesthesia and mechanical ventilation are performed annually. Postoperative pulmonary complications (PPCs) significantly impact clinical outcomes, increasing morbidity and hospitalization duration. Cohort studies have reported a 20-30% risk of PPCs in patients undergoing general anesthesia. Protective ventilation strategies, including low tidal volumes (6-8 mL/kg predicted body weight) and positive end-expiratory pressure (PEEP), have shown to reduce PPCs. However, high tidal volumes (10-15 mL/kg) remain prevalent in routine practice.

The "RuVent-A" study will collect data on respiratory support methodologies, initial ventilation parameters, types of surgical interventions, and associated PPC rates in the Russian Federation. This observational study will analyze patient and equipment data across participating centers without altering routine clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years undergoing surgical procedures with general anesthesia and respiratory support.

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients (aged ≥18 years) undergoing surgical procedures under general anesthesia with respiratory support in participating medical centers across the Russian Federation. The study will focus on a wide range of surgical specialties, including but not limited to general surgery, orthopedics, neurosurgery, vascular surgery, and thoracic surgery.
  Patients with various comorbidities (e.g., obesity, chronic obstructive pulmonary disease, smoking, sleep apnea) that may influence respiratory support strategies will be included to provide a comprehensive assessment of perioperative respiratory management and its outcomes.
  No specific exclusion criteria will be applied, allowing for the inclusion of a diverse and representative cohort of surgical patients.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-05-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Pulmonary Complications (PPCs) | 30 days after surgery
  The frequency of postoperative pulmonary complications (PPCs) will be measured, including conditions such as atelectasis, hypoxemia, pneumonia, acute respiratory distress syndrome (ARDS), and bronchospasm. PPCs will be evaluated based on clinical and diagnostic criteria following surgery.

SECONDARY OUTCOMES:
Level of end-expiratory pressure during anesthesia | During surgery (intraoperative period).
  The level of end-expiratory pressure during anesthesia used by the anesthesiologist will be assessed
Use of Alveolar Recruitment Maneuvers During Anesthesia | During surgery (intraoperative period).
  The frequency of alveolar recruitment maneuvers used during general anesthesia will be assessed.
Frequency of Non-Invasive Ventilation and High-Flow Oxygen Therapy Post-Extubation | 30 days after surgery
  The frequency of non-invasive ventilation (NIV) and high-flow oxygen therapy (HFOT) applied after extubation will be evaluated to determine their role in preventing PPCs.
Duration of Intraoperative and Postoperative Mechanical Ventilation | Intraoperative and up to 24 hours postoperatively.
  Duration of Intraoperative and Postoperative Mechanical Ventilation
Incidence of Hypoxemia Post-Surgery | 30 days after surgery
  The occurrence of hypoxemia (SpO2 <92%) after surgery will be documented, along with the requirement for oxygen therapy.
Level of inspiratory oxygen fraction during anesthesia | During surgery (intraoperative period).
  The level of inspiratory oxygen fraction during anesthesia used by the anesthesiologist will be assessed
Level of tidal volume during anesthesia | During surgery (intraoperative period).
  The level of tidal during anesthesia used by the anesthesiologist will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Yaroshetskiy, MD, Principal Investigator — Sechenov First Moscow State Medical University

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) Sharing Statement
  Individual participant data (IPD) will not be shared due to the following reasons:
  Privacy and Confidentiality: The study involves sensitive patient data, and ensuring patient confidentiality is a top priority. Although the data will be anonymized, sharing IPD could still pose risks of re-identification.
  Regulatory and Ethical Considerations: Sharing IPD may not comply with local regulations and ethical guidelines governing patient data use in the Russian Federation.
  Study Scope: The primary objective of this study is to analyze aggregated data to inform clinical practices rather than to enable secondary analyses or external collaborations.